CLINICAL TRIAL: NCT00968747
Title: The Effect of Acute Nutritional Challenges on FGF21 Levels in Humans
Brief Title: Regulation of FGF21 by Nutritional Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jody Dushay, MD, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009P-000073
Record Dates: First submitted 2009-07-31; First posted 2009-08-31 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fasting; Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Fasting; Fast; healthy; diet; study; manipulation; dietary; FGF21; Fibroblast growth factor; PTRF; Polymerase 1 and transcript release factor; adipose; fat; blood; inpatient; outpatient; NAFLD; metabolism
MeSH Terms: conditions — Fasting; Non-alcoholic Fatty Liver Disease; Platelet Glycoprotein IV Deficiency | interventions — Angptl4 protein, mouse; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fasting (Healthy). (Experimental): Participants will fast for 72 hours during an inpatient stay at the Beth Israel Deaconess Medical Center in Boston, MA. Blood samples will be collected daily and two fat samples will be obtained by a trained surgeon. (We are no longer recruiting for Study Arm A).
  Interventions: Behavioral: Fasting
- Fasting (NAFLD) (Experimental): Participants with liver-biopsy diagnosed non-alcoholic fatty liver disease (NAFLD) will fast for 72 hours during an inpatient stay at the Beth Israel Deaconess Medical Center in Boston, MA. Blood samples will be collected daily, and participants will have an MRI before and after the fast.
  Interventions: Behavioral: Fasting
- Hypocaloric diet (NAFLD) (Experimental): Participants will follow a low-calorie diet until they lose 3-5% of their body weight. Participants will have weekly outpatient visits at Beth Israel Deaconess Medical Center in Boston, MA for weight measurements. Participants will have blood drawn before and after the diet. Participants will also have an MRI before and after the diet.
  Interventions: Behavioral: Diet
- Oral carbohydrate challenge (Experimental): Participants will fast for 16 hours overnight then ingest drinks containing fructose, glucose or a mixture of fructose and glucose. Blood will be drawn postprandially at specified timepoints for up to 5 hours
  Interventions: Dietary Supplement: oral carbohydrate challenge

INTERVENTIONS:
Behavioral: Fasting — Participants will fast for 72 hours and may consume only water and vitamins.
  Arms: Fasting (Healthy).
Behavioral: Fasting — Participants will fast for 72 hours and may consume only water and vitamins.
  Arms: Fasting (Healthy).; Fasting (NAFLD)
Behavioral: Diet — Participants will follow a low-calorie diet until they lose 3-5% of their body weight.
  Arms: Hypocaloric diet (NAFLD)
Dietary Supplement: oral carbohydrate challenge — Participants will fast for 16 hours and then drink a beverage containing glucose, fructose or a mixture of both
  Arms: Oral carbohydrate challenge

SUMMARY:
The purpose of this study is to examine how acute nutritional challenges affect levels of several proteins involved in metabolism. These proteins will be measured in blood and fat tissue.

This study will have several aims.

One aim is to examine the effect of 72 hours of fasting on fibroblast growth factor-21 (FGF-21) levels. Participants will spend 3 days and nights in the Clinical Research Center at the Beth Israel Deaconess Medical Center in Boston, MA. Daily blood samples will be taken. Two fat samples will be taken prior to and at the end of the fast. A subset of participants will also have two MRIs, one prior to and one at the end of the fast. We will study healthy adults and obese adults with liver-biopsy-diagnosed non-alcoholic fatty liver disease (NAFLD). THIS STUDY ARM IS CURRENTLY NOT RECRUITING

Another aim is to examine the effect of low-calorie diet on FGF-21 levels. Subjects will follow a hypocaloric diet that will be designed to achieve 3-5% weight loss. We will enroll participants with liver-biopsy-diagnosed non-alcoholic fatty liver disease. Participants will report weekly to the Clinical Research Center at Beth Israel Deaconess Medical Center for weight measurements. Blood will be drawn before and after the weight loss. Participants will also have an MRI before and after the weight loss.

THIS ARM IS CURRENTLY NOT RECRUITING

Another aim of the study is to examine the effect of acute ingestion of glucose, fructose, and other sugars on serum FGF21 levels. Subjects in this study will be lean volunteers and individuals with metabolic syndrome.

THIS ARM IS CURRENTLY RECRUITING

DETAILED DESCRIPTION:
Participation in this study involves fasting overnight, drinking a sweet beverage, and several blood draws through an IV line. Each subject may drink up to 5 different sweet beverages, separated by 2 weeks.

ELIGIBILITY:
72-hour fast in healthy volunteers (Study Arm A):

Inclusion Criteria:

* Age 18-50 years
* Body Mass Index 21-26 kg/m^2
* Ability to give informed consent
* Ability to follow verbal and written instructions in English

Exclusion Criteria:

* Type 1 or Type 2 diabetes mellitus diagnosed according to the American Diabetes Association criteria
* Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure)
* Tobacco, marijuana, or intravenous drug use within 1 year of screening visit
* Recent weight change (>3 kg within 6 months of screening visit)
* Malignancy treated with chemotherapy within past 3 years
* History of depression, psychosis, or other psychiatric illness requiring hospitalization
* History of hyperthyroidism
* Renal insufficiency (creatinine clearance < 50 ml/min)
* Transaminases > 2X above the normal range
* Known liver disease
* Pregnancy within 12 months of screening visit
* Lactation within 12 months of screening visit
* Failure to use medically approved contraceptive methods (oral contraceptive, 2 barrier methods, surgical sterilization)
* History of an eating disorder (anorexia, bulimia, or laxative abuse)
* History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
* New diagnosis of hypothyroidism within 1 year of screening visit or change in dose of thyroid hormone within 3 months of screening visit
* History of alcohol abuse within the past 3 years
* History of keloid formation
* History of allergy to lidocaine or marcaine
* Use of plavix, coumadin, or heparin

  72-hour fast or hypocaloric diet in subjects with non-alcoholic fatty liver disease (NAFLD) (Study Arms B & C):

Inclusion Criteria:

* Age 18-60
* BMI 25-45 kg/m^2
* Known nonalcoholic fatty liver disease based on liver biopsy
* Ability to give informed consent
* Ability to follow verbal and written instructions in English

Exclusion Criteria:

* Type I diabetes mellitus diagnosed according to the American Diabetes Association criteria or Type II diabetes mellitus with A1c > 7.5% or taking metformin or thiazolidinediones
* Coronary Heart Disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure)
* Uncontrolled hypertension (BP > 150/90 mmHg on or off antihypertensive medication)
* Tobacco, marijuana, or intravenous drug use within 1 year of screening visit
* Recent weight change (> 3 kg within 6 months of screening visit)
* Malignancy treated with chemotherapy within the past 3 years
* History of depression, psychosis, or other psychiatric illness requiring hospitalization
* History of hypo or hyperthyroidism
* Renal insufficiency (creatinine clearance < 50 ml/min)
* Pregnancy within 12 months of screening visit
* Lactation within 12 months of screening visit
* Failure to use medically approved contraceptive methods (oral contraceptive, 2 barrier methods, surgical sterilization)
* History of an eating disorder (anorexia, bulimia, or laxative abuse)
* History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
* New diagnosis of hypo or hyperthyroidism within 1 year of screening visit or change in dose of thyroid hormone within 3 months of screening visit
* History of alcohol abuse within the past 3 years
* Cardiac pacemaker or aneurysm clips
* Metal implants in the body (pins, plates, shrapnel, intact bullets, IUD)
* Claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Fibroblast Growth Factor 21 levels in serum and fat | before and after dietary intervention
  Change in FGF21 levels following nutritional intervention.

SECONDARY OUTCOMES:
Polymerase 1 and Transcript Release Factor levels in fat | Prior to fasting and at the end of the 72-hour fast in healthy participants and participants with NAFLD
Urine and serum ketosis | Daily during the 72-hour fast for healthy participants and participants with NAFLD
Hepatic fat content | Before and after the 72-hour fast or hypocaloric diet in participants with NAFLD
change in serum triglyceride levels | following fructose and glucose ingestion
change in glucose and insulin levels | following fructose and glucose ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Jody Dushay, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States